CLINICAL TRIAL: NCT04831762
Title: MARQUEURS DE DEVELOPPEMENT DE L'ATTENTION EXECUTIVE CHEZ L'ENFANT : POPULATIONS VARIEES
Brief Title: Markers of Executive Attention Development in Preschoolers - Behavioral Measures in Various Populations
Acronym: MEDiATE-PRV
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A03209-30
Record Dates: First submitted 2021-04-02; First posted 2021-04-05 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-03

CONDITIONS: Attention Deficit
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Attention Network task (computerized) — Computer-based game challenging orienting and executive attention. The subject must chose which side an animal is going, using left and right buttons, depending on the validity of a cue and the congruency of flankers.
  Other Names: Child ANT, flankers task
Behavioral: Head-toes-knees-schoulders — Following motor commands such as touch your head when they are congruent or incongruent.
  Other Names: HTKS
Behavioral: Laby 5-12 — Test of motor planning using labyrinths
Behavioral: M-ABC 2 — Test of motor functions using various subtests of gross and fine motor function.
Behavioral: Stroop animals — Stroop test for preK children using animals instead of words

SUMMARY:
Executive attention is essential for emotional and behavioral self-regulation. There is inter-individual variability in the level of efficiency of executive attention from kindergarten entry, and this variability predicts children's academic performance at entry to elementary school and beyond. It is therefore essential to better understand the early stages of executive attention development and self-regulation from an early age in order to develop tools for early detection of executive attention disorders, so that school accommodations can be proposed as early as possible.

In previous work, we have identified early tactile information processing skills that underpin the development of executive attention. We would like to extend this work to a diverse population of preschool children, in order to consider new tools for the early detection of attention disorders. The MEDiATE-PRV project aims to compare the performance obtained in a validated attentional task in preschool children with assessments of tactile information processing, in relation to the psychomotor and executive development of the child. We will include 200 children aged 4 years to 5 years 11 months with different risk factors for ADHD.

ELIGIBILITY:
Inclusion Criteria:

* Attending preschool
* Parental informed consent

Exclusion Criteria:

- None

Ages: 48 Months to 71 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preschoolers 48 to 71 months of age.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-10-01 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
ANT performance | 48 to 71 months of age
  Reaction time in ms to ANT trials with a correct answer
Tactile processing score | 48 to 71 months of age
  Score to the sensory profile tactile subtest

CONTACTS AND LOCATIONS:
Locations (1):
- Comete U1075 Inserm Unicaen, Caen, France